CLINICAL TRIAL: NCT03335007
Title: Pretreatment Aceclofenac Effect on Pain and Analgesic Intake After Endodontic Treatment: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Pretreatment Aceclofenac Effect on Pain and Analgesic Intake After Endodontic Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermeen AwadAllah Abbas Ibrahim, Principal Investigator, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEBD-CU-2015-5-146
Record Dates: First submitted 2017-10-29; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Aceclofenac; pain; irreversible pulpitis
MeSH Terms: conditions — Pain | interventions — aceclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aceclofenac (Experimental): Aceclofenac 100 mg tablet
  Interventions: Drug: Aceclofenac
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aceclofenac — Aceclofenac 100 mg tablet given one hour before starting the root canal treatment
  Other Names: Bristaflam
  Arms: Aceclofenac
Other: Placebo — Placebo tablet given one hour before starting the root canal treatment
  Arms: Placebo

SUMMARY:
The aim of this prospective, randomized, double-blind, clinical trial is to evaluate the effect of a preoperative, single, oral dose of aceclofenac (100 mg) on postendodontic pain at 6, 24 and 48 hours, postoperative pain at injection area at 6, 24 and 48 hours and analgesic intake after single-visit root canal treatment.

DETAILED DESCRIPTION:
* Patients will be clinically and radiographically examined and their eligibility will be assessed and preoperative pain will be measured using Heft-Parker VAS. Eligible patients will be treated in one visit.
* Patients will be randomly assigned to one of 2 groups: experimental group (taking a 100 mg of Aceclofenac) and the control group (taking a placebo tablet). Each tablet will be taken one hour before the initiation of single-visit endodontic therapy. Each participant will receive a standard inferior alveolar nerve block injection of 1.8 ml of 2% mepivacaine with 1:100,000 epinephrine. After endodontic treatment, patients will be given postoperative instructions and informed, in case of pain, to receive ibuprofen 200 mg as rescue medication.
* Postendodontic pain intensity and incidence at the different pain categories (No, mild, moderate, severe) will be assessed 6, 24, and 48 hours postoperatively using Heft-Parker visual analogue scale (HP-VAS). Postoperative pain at injection area will be assessed at 6,24 and 48 hours using HP-VAS. Analgesic intake throughout the 48 hours will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good health (American Society of Anesthesiologists Class I or Class II).
* Patients having symptomatic irreversible pulpitis in one of their mandibular molars
* Age is 18 years or older.
* Patients who can understand Heft- Parker Visual Analogue Scales.
* Patients able to sign informed consent.

Exclusion Criteria:

* Patients allergic to aceclofenac or Mepivacaine.
* Pregnant or nursing women.
* Patients having active pain in more than one molar in the same quadrant.
* Administration of analgesics within 12 h before the administration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Postendodontic pain rate change | At 6, 24 and 48 hours after root canal treatment.
  Postendodontic pain will be measured using Heft-Parker visual analogue scale. No or mild pain response will be considered success.

SECONDARY OUTCOMES:
Postoperative pain at injection area | At 6, 24 and 48 hours after root canal treatment.
  Postoperative pain at injection area will be measured with Heft-Parker visual analogue scale. No or mild pain response will be considered success.
Analgesic intake | Within 48 hours after single root canal treatment.
  Incidence of analgesic intake

CONTACTS AND LOCATIONS:
Overall Officials: Nermeen A Abbas, Postgraduate, Principal Investigator — Cairo University; Suzan AW Amin, PhD, Study Director — Cairo University; Shaimaa Gawdat, PhD, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Praveen R, Thakur S, Kirthiga M. Comparative Evaluation of Premedication with Ketorolac and Prednisolone on Postendodontic Pain: A Double-blind Randomized Controlled Trial. J Endod. 2017 May;43(5):667-673. doi: 10.1016/j.joen.2016.12.012. Epub 2017 Mar 17. PMID 28320541
- [Background] Attar S, Bowles WR, Baisden MK, Hodges JS, McClanahan SB. Evaluation of pretreatment analgesia and endodontic treatment for postoperative endodontic pain. J Endod. 2008 Jun;34(6):652-5. doi: 10.1016/j.joen.2008.02.017. Epub 2008 Apr 2. PMID 18498882